CLINICAL TRIAL: NCT02650401
Title: A Phase 1/2, Open-Label, Dose-Escalation And Expansion Study Of Entrectinib (Rxdx-101) In Pediatrics With Locally Advanced Or Metastatic Solid Or Primary CNS Tumors And/Or Who Have No Satisfactory Treatment Options
Brief Title: Study Of Entrectinib (Rxdx-101) in Children and Adolescents With Locally Advanced Or Metastatic Solid Or Primary CNS Tumors And/Or Who Have No Satisfactory Treatment Options
Acronym: STARTRK-NG
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXDX-101-03; CO40778 (Other: Hoffmann-La Roche); 2023-505088-35-00 (EU CTIS Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-08 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors; CNS Tumors
Keywords: TRK; Tyrosine kinase; NTRK; NTRK1; NTRK2; NTRK3; ROS1; ALK; Pediatric; Relapsed; Refractory; Solid Tumor; Metastatic Cancer; Gene rearrangement; Neuroblastoma; Infantile fibrosarcoma; Secretory breast cancer; Congenital mesoblastic nephroma; Pontine glioma; Brain tumors; CNS tumors; Sarcoma; Ewing sarcoma; Glial tumors; Salivary Gland Cancer (MASC); Papillary thyroid cancer; Medulloblastoma; Wilms tumor (anaplastic)
MeSH Terms: conditions — Central Nervous System Neoplasms; Recurrence; Neoplasm Metastasis; Neuroblastoma; Nephroma, Mesoblastic; Brain Neoplasms; Sarcoma; Sarcoma, Ewing; Glioma; Salivary Gland Neoplasms; Thyroid Cancer, Papillary; Medulloblastoma; Wilms Tumor | interventions — entrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Extracranial solid tumors harboring NTRK1/2/3, (Active Comparator): Arm closed for further enrollment
  ROS1, ALK non-gene fusion molecular alterations
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- CNS tumors harboring- NTRK1/2/3, ROS1, ALK (Active Comparator): Arm closed for further enrollment
  molecular alterations, including gene fusions
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- Neuroblastoma (Active Comparator): Arm closed for further enrollment
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- Non-neuroblastoma, extracranial solid tumors (Active Comparator): Arm closed for further enrollment
  harboring - NTRK1/2/3, ROS1, ALK gene fusions
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- Any participant unable to swallow capsules (Active Comparator): Arm closed for further enrollment
  Any participant who otherwise meet all other eligibility criteria
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- Expansion: CNS tumors harboring NTRK1/2/3, ROS1 (Active Comparator): gene fusions
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib
- Expansion: Extracranial solid tumors harboring NTRK1/2/3, ROS1 (Active Comparator): NTRK 1,2,3 and ROS1 fusions
  Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib

INTERVENTIONS:
Drug: Entrectinib — TRKA/B/C, ROS1, and ALK inhibitor
  Other Names: RXDX-101

SUMMARY:
This is an open-label, Phase 1/2 multicenter dose escalation study in pediatric patients with relapsed or refractory extracranial solid tumors (Phase 1), with additional expansion cohorts (Phase 2) in patients with primary brain tumors harboring NTRK1/2/3 or ROS1 gene fusions, and extracranial solid tumors harboring NTRK1/2/3 or ROS1 gene fusions.

ELIGIBILITY:
Inclusion Criteria:

1. Disease status:

   * Phase 1 portion (closed): Participants must have measurable or evaluable disease, as defined by RECIST v1.1
   * Phase 2 portion:

     * Part B: Participants must have measurable or evaluable disease, as defined by RANO
     * Part C (closed): Participants must have measurable or evaluable disease, as defined by RECIST v1.1 ± Curie Scale
     * Part D: Participants must have measurable or evaluable disease, as defined by RECIST v1.1
     * Part E (closed): Participants must have measurable or evaluable disease, as defined by RECIST v1.1 ± Curie Scale or RANO
2. Tumor type:

   * Phase 1 portion:

     * Part A: Relapsed or refractory extracranial solid tumors
   * Phase 2 portion

     * Part B: Primary brain tumors with NTRK1/2/3 or ROS1 gene fusions; gene fusions are defined as those predicted to translate into a fusion protein with a functional TRKA/B/C or ROS1 kinase domain, without a concomitant second oncodriver as determined by a nucleic acid-based diagnostic testing method
     * Part D: Extracranial solid tumors (including NB) with NTRK1/2/3 or ROS1 gene fusions; gene fusions are defined as those predicted to translate into a fusion protein with a functional TRKA/B/C or ROS1 kinase domain, without a concomitant second oncodriver as determined by a nucleic acid-based diagnostic testing method
3. Histologic/molecular diagnosis of malignancy at diagnosis or the time of relapse
4. Archival tumor tissue from diagnosis or, preferably, at relapse
5. Performance status: Lansky or Karnofsky score ≥ 60% and minimum life expectancy of at least 4 weeks
6. Prior therapy: Participants must have a disease that is locally advanced, metastatic, or where surgical resection is likely to result in severe morbidity, and who have no satisfactory treatment options for solid tumors and primary CNS tumors that are neurotrophic tyrosine receptor kinase (NTRK) or ROS1 fusion-positive
7. Participants must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to enrollment
8. Adequate organ and neurologic function
9. Females of childbearing potential must have a negative serum pregnancy test during screening and be neither breastfeeding nor intending to become pregnant during study participation. Agreement to remain abstinent or use use combined contraceptive methods prior to study entry, for the duration of study participation and in the following 90 days after discontinuation of study treatment.
10. For male participants with a female partner of childbearing potential or a pregnant female partner: Agreement to remain abstinent or use a condom during the treatment period and for at least 3 months after the last dose of study drug

Exclusion Criteria:

1. Receiving other experimental therapy
2. Known congenital long QT syndrome
3. History of recent (3 months) symptomatic congestive heart failure or ejection fraction ≤50% at screening
4. Known active infections
5. Familial or personal history of congenital bone disorders, bone metabolism alterations or osteopenia
6. Receiving Enzyme Inducing Antiepileptic Drugs (EIAEDs) within 14 days of first dose.
7. Prior treatment with approved or investigational TRK or ROS1 inhibitors
8. Known hypersensitivity to entrectinib or any of the other excipients of the investigational medicinal product
9. Patients with NB with bone marrow space-only disease
10. Incomplete recovery from acute effects of any surgery prior to treatment.
11. Active gastrointestinal disease or other malabsorption syndromes that would impact drug absorption.
12. Other severe acute or chronic medical or psychiatric condition or lab abnormality that may increase the risk associated with study participation, drug administration or may interfere with the interpretation of study results.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Approximately 6 months
  Assessed by National Cancer Institute Common Terminology for Adverse Events Criteria (NCI CTCAE v4.03)
Recommended Phase 2 Dose (RP2D) of F1 Formulation In Pediatric Participants Able To Swallow Intact Capsules | Approximately 6 months
  Assessed by NCI CTCAE v4.03
Recommended Phase 2 Dose (RP2D) of F06 Formulation In Pediatric Participants Able To Swallow Intact Capsules | Approximately 6 months
  Assessed by NCI CTCAE v4.03
Recommended Phase 2 Dose (RP2D) of F06 Formulation In Pediatric In Participants Dosed Via Feeding Tube (Nasogastric Tube Or Gastric Tube) | Approximately 6 months
  Assessed by NCI CTCAE v4.03
Recommended Phase 2 Dose (RP2D) Of Minitablets/F15 Formulation In Pediatric Participants Unable To Swallow Intact Capsules | Approximately 6 months
  Assessed by NCI CTCAE v4.03
Cohort B: Objective Response Rate (ORR) | Approximately 6 months
  Assessed by RANO per the BICR
Cohort D: ORR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR

SECONDARY OUTCOMES:
Safety and Tolerability - AE, ECG and Labs assessed by NCI CTCAE v4.03 | Approximately 24 months
  AE, ECG and Labs assessed by NCI CTCAE v4.03
Maximum observed plasma drug concentration (Cmax) using F1 Formulation | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Maximum observed plasma drug concentration (Cmax) using F06 Formulation given intact | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Maximum observed plasma drug concentration (Cmax) using F06 Formulation administered via feeding tube | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Maximum observed plasma drug concentration (Cmax) using minitablets/F15 | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Time to Cmax, by inspection (Tmax) using F1 Formulation | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Time to Cmax, by inspection (Tmax) using F06 Formulation given intact | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Time to Cmax, by inspection (Tmax) using F06 Formulation administered via feeding tube | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Time to Cmax, by inspection (Tmax) using minitablets/F15 | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
AUC at steady state (AUCss) using F1 Formulation | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
AUC at steady state (AUCss) using F06 Formulation given intact | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
AUC at steady state (AUCss) using F06 Formulation administered via feeding tube | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
AUC at steady state (AUCss) using minitablets/F15 | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Terminal half life (t½) using F1 Formulation | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Terminal half life (t½) using F06 Formulation given intact | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Terminal half life (t½) using F06 Formulation administered via feeding tube | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Terminal half life (t½) using minitablets/F15 | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Area under the drug concentration by time curve (AUC) using F1 Formulation | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Area under the drug concentration by time curve (AUC) using F06 Formulation given intact | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Area under the drug concentration by time curve (AUC) using F06 Formulation administered via feeding tube | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Area under the drug concentration by time curve (AUC) using minitablets/F15 | Approximately 24 months
  Assessed by plasma concentrations obtained on Days 1, 2, 8, 15, 22 (Cycle 1), Days 1, 2 (Cycle 2) and on Day 1 of every cycle thereafter
Cohort A, D, or E: Clinical Benefit Rate (CBR) | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Cohort B or E: CBR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Cohort C: CBR | Approximately 6 months
  Assessed by the Curie scale per the BICR and investigator
Cohort A, D, or E: Progression-free Survival (PFS) | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Cohort B or E: PFS | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Cohort C: PFS | Approximately 6 months
  Assessed by the Curie scale per the BICR and investigator
Cohort A, D, or E: Overall Survival (OS) | Approximately 6 months
  Assessed by RECIST v1.1
Cohort B or E: OS | Approximately 6 months
  Assessed by RANO
Cohort A, D, or E: ORR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Cohort B or E: ORR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Cohort C: ORR | Approximately 6 months
  Assessed by the Curie scale per the BICR and investigator
Cohort A, D, or E: Time to response (TTR) | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Cohort B or E: TTR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Cohort C: TTR | Approximately 6 months
  Assessed by the Curie scale per the BICR and investigator
Cohort A, D, or E: Duration of Response (DOR) | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Cohort B or E: DOR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Cohort C: DOR | Approximately 6 months
  Assessed by the Curie scale per the BICR and investigator
Phase 2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort B or E): ORR | Approximately 6 months
  Assessed by RANO per the investigator
Phase 2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort D or E): ORR | Approximately 6 months
  Assessed by RECIST v1.1 per the investigator
Phase 1/2 Participants with NTRK1/2/3 gene fusions (Cohort A, D, or E): ORR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 gene fusions (Cohort B or E): ORR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 1/2 Participants with ROS1 gene fusions (Cohort A, D, or E): ORR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with ROS1 gene fusions (Cohort B or E): ORR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort A, D, or E): ORR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort B or E): ORR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort B or E): DOR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort D or E): DOR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 gene fusions (Cohort A, D, or E): DOR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 gene fusions (Cohort B or E): DOR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 1/2 Participants with ROS1 gene fusions (Cohort A, D, or E): DOR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with ROS1 gene fusions (Cohort B or E): DOR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort A, D, or E): DOR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort B or E): DOR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort B or E): TTR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort D or E): TTR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 gene fusions (Cohort A, D, or E): TTR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 gene fusions (Cohort B or E): TTR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 1/2 Participants with ROS1 gene fusions (Cohort A, D, or E): TTR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with ROS1 gene fusions (Cohort B or E): TTR | Approximately 6 months
  Assessed by RANO per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort A, D, or E): TTR | Approximately 6 months
  Assessed by RECIST v1.1 per the BICR and investigator
Phase 1/2 Participants with NTRK1/2/3 or ROS1 gene fusions (Cohort B or E): TTR | Approximately 6 months
  Assessed by RANO per the BICR and investigator

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- United States (15):
  - University of California San Diego, La Jolla, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Egleston Children's Hospital at Emory University Atlanta, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University,St. Louis Children's Hospital, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science Uni, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children'S Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer and Hematology Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
- The Hospital for Sick Children, Toronto, Ontario, Canada
- China (2):
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Beijing Children's Hospital, Capital Medical University, Beijing
- France (2):
  - Centre Leon Berard, Lyon
  - Hôpital de la Timone, Oncologie Pédiatrique, Marseille
- Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg, Germany
- Hong Kong Children's Hospital, Hong Kong, Hong Kong
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- Hospital Infantil Universitario Nino Jesus, Madrid, Spain
- United Kingdom (2):
  - Royal Marsden Hospital (Sutton), London
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing.

REFERENCES:
- [Derived] Desai AV, Bagchi A, Armstrong AE, van Tilburg CM, Basu EM, Robinson GW, Wang H, Casanova M, Andre N, Campbell-Hewson Q, Wu Y, Cardenas A, Ci B, Ryklansky C, Devlin CE, Meneses-Lorente G, Wulff J, Hutchinson KE, Gajjar A, Fox E. Efficacy and safety of entrectinib in children with extracranial solid or central nervous system (CNS) tumours harbouring NTRK or ROS1 fusions. Eur J Cancer. 2025 May 2;220:115308. doi: 10.1016/j.ejca.2025.115308. Epub 2025 Feb 22. PMID 40086048
- [Derived] Desai AV, Robinson GW, Gauvain K, Basu EM, Macy ME, Maese L, Whipple NS, Sabnis AJ, Foster JH, Shusterman S, Yoon J, Weiss BD, Abdelbaki MS, Armstrong AE, Cash T, Pratilas CA, Corradini N, Marshall LV, Farid-Kapadia M, Chohan S, Devlin C, Meneses-Lorente G, Cardenas A, Hutchinson KE, Bergthold G, Caron H, Chow Maneval E, Gajjar A, Fox E. Entrectinib in children and young adults with solid or primary CNS tumors harboring NTRK, ROS1, or ALK aberrations (STARTRK-NG). Neuro Oncol. 2022 Oct 3;24(10):1776-1789. doi: 10.1093/neuonc/noac087. PMID 35395680
- [Derived] Doebele RC, Drilon A, Paz-Ares L, Siena S, Shaw AT, Farago AF, Blakely CM, Seto T, Cho BC, Tosi D, Besse B, Chawla SP, Bazhenova L, Krauss JC, Chae YK, Barve M, Garrido-Laguna I, Liu SV, Conkling P, John T, Fakih M, Sigal D, Loong HH, Buchschacher GL Jr, Garrido P, Nieva J, Steuer C, Overbeck TR, Bowles DW, Fox E, Riehl T, Chow-Maneval E, Simmons B, Cui N, Johnson A, Eng S, Wilson TR, Demetri GD; trial investigators. Entrectinib in patients with advanced or metastatic NTRK fusion-positive solid tumours: integrated analysis of three phase 1-2 trials. Lancet Oncol. 2020 Feb;21(2):271-282. doi: 10.1016/S1470-2045(19)30691-6. Epub 2019 Dec 11. PMID 31838007